CLINICAL TRIAL: NCT06681506
Title: A New Cardiac Rehabilitation Treatment in the Application of Ischemic Heart Disease: a Prospective, Randomized Controlled Clinical Study
Brief Title: A New Cardiac Rehabilitation Treatment in the Application of Ischemic Heart Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government)
Responsible Party: Principal Investigator, Ya-Wei Xu, Chief Physician, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rehabilitation-ICM
Record Dates: First submitted 2024-11-03; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Ischemic Heart Disease; Cardiac Rehabilitation
Keywords: coronary atherosclerotic cardiopathy; Cardiac Shock Wave Therapy; exercise rehabilitation; cardiac rehabilitation; Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia | interventions — Exercise Therapy; Counterpulsation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The new rehabilitation group (Experimental): Routine drug therapy + new cardiac rehabilitation therapy, a new cardiac rehabilitation treatment reference guide requirements, according to the actual circumstance of patients treated with 1-3 months intervention.
  Interventions: Device: Metronomic breathing, exercise rehabilitation, external counterpulsation, extracorporeal shock wave.
- The traditional rehabilitation group. (Active Comparator): Routine drug therapy + traditional cardiac rehabilitation therapy, traditional cardiac rehabilitation treatment for reference domestic and international guidelines and consensus, according to the actual circumstance of patients treated with 1-3 months intervention.
  Interventions: Device: bedside rehabilitation and breathing, balance, flexibility, movement rehabilitation

INTERVENTIONS:
Device: Metronomic breathing, exercise rehabilitation, external counterpulsation, extracorporeal shock wave. — Phase I rehabilitation(Metronomic breathing，exercise rehabilitation）,Phase II rehabilitation (exercise rehabilitation, external counterpulsation, extracorporeal shock) wave.)
  Arms: The new rehabilitation group
Device: bedside rehabilitation and breathing, balance, flexibility, movement rehabilitation — Phase I rehabilitation (bedside rehabilitation, breathing rehabilitation), Phase II rehabilitation (breathing, balance, flexibility, movement)
  Arms: The traditional rehabilitation group.

SUMMARY:
Cardiac rehabilitation is an important link in cardiovascular disease. This study mainly explores the effectiveness of new cardiac rehabilitation therapy (early respiratory rehabilitation, phase I rehabilitation, exercise therapy, external counterpulsation, extracorporeal shock wave, etc.) on patients with ischemic heart disease such as coronary heart disease and heart failure, and the compliance of home rehabilitation compared with traditional cardiac rehabilitation therapy (traditional exercise rehabilitation, rehabilitation education, etc.).

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled study, follow the principle of PICOST design, specific as follows: Participants (the list) : preliminary clinical diagnosis of coronary atherosclerotic heart disease, heart failure. Intervention (Intervention) : conventional drug therapy + new cardiac rehabilitation therapy, a new cardiac rehabilitation treatment reference guide requirements, according to the actual circumstance of patients treated with 1-3 months Intervention. Comparator(control): conventional drug therapy + traditional cardiac rehabilitation therapy. The traditional cardiac rehabilitation therapy referred to domestic and international guidelines and consensus, and used 1 week-3 months of treatment intervention according to the actual situation of patients. Outcome (the end) : the primary end point: D_SPECT examination, were followed up for 6 months to evaluate myocardial perfusion imaging is reduce ischemic area. The secondary end point: 1) the blood biochemical examination and myocardial necrosis markers, etc.; 2) the cardiopulmonary exercise testing: maximum kilograms oxygen uptake and anaerobic threshold when the maximum kilograms oxygen uptake; 3) the major adverse cardiovascular events: cardioascular death, non-fatal myocardial infarction, unplanned coronary artery reconstruction, stroke, heart failure and angina associated hospitalized again; 4) patients family rehabilitation treatment adherence

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 85 years old
* Female subjects no pregnancy
* The main admission diagnosis of ischemic heart disease (coronary heart disease, myocardial infarction, ischemic heart failure, etc.)
* The need for cardiac rehabilitation treatment

Exclusion Criteria:

* acute respiratory distress syndrome (ARDS);
* acute episode of COPD;
* uncontrolled pulmonary infection;
* acute heart failure; acute pulmonary embolism;
* acute myocarditis/pericarditis;
* severe arrhythmia (degree II or III atrioventricular block, atrial flutter, or atrial fibrillation);
* sternotomy, rib fracture, thoracic deformity, or other neurological diseases that may affect respiratory muscles

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline myocardial infarct area at 6 months | 1 day of inclusions and 6 months after the first treatment.
  The location and extent of myocardial infarction were determined by D-SPECT.

SECONDARY OUTCOMES:
6 months hemodynamic changes in relative to the baseline | 1 day of inclusions and 6 months after the first treatment.
  Noninvasive hemodynamic evaluation of hemodynamic state, such as, the larger the value of Stroke volume, Stroke volume index, Cardiac output, Cardiac output index parameters, the smaller the value of Systemic vascular resistance, Systemic vascular resistance index parameters, the better the function of the patient's heart and arterial vessels.
Change from baseline peak oxygen consumption at 6 months | 1 day of inclusions and 6 months after the first treatment.
  maximum oxygen and maximum kilogram oxygen uptake accessed during Cardiopulmonary Exercise Testing (CPET)

OTHER OUTCOMES:
Major adverse cardiovascular events (MACE） | From the date of inclusion until the date of documented adverse events with 6 months
  cardiovascular death, non-fatal myocardial infarction, unplanned coronary revascularization, stroke, heart failure, and angina-related rehospitalization
Other treatment-related adverse reactions | From the date of inclusion until the date of treatment-related adverse reactions within 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes